CLINICAL TRIAL: NCT01504464
Title: Evaluation the Effects of Intra-articular Injection of Mesenchymal Stem Cells in Patients With Knee Joint Osteoarthritis, Triple Blind Randomized Clinical Trial
Brief Title: The Effects of Intra-articular Injection of Mesenchymal Stem Cells in Knee Joint Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Royan-Bone-010
Record Dates: First submitted 2012-01-03; First posted 2012-01-05 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis
Keywords: knee joint osteoarthritis mesenchymal stem cell
MeSH Terms: conditions — Osteoarthritis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mesenchymal stem cell (Experimental): Patients with knee joint osteoarthritis who underwent intra articular mesenchymal stem cell injection.
  Interventions: Biological: mesenchymal stem cell
- placebo (Experimental): The patients who are in control group and underwent placebo injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mesenchymal stem cell — intra articular injection of mesenchymal stem cell
  Other Names: stem cell transplantation
  Arms: mesenchymal stem cell
Biological: Placebo — Patients with knee joint osteoarthritis who underwent intra articular placebo injection
  Arms: placebo

SUMMARY:
Osteoarthritis of the knee is one of the most common causes of disability among elderly. As the disease progresses the cartilage become frustrated, surrounding bone react to become thicker and inflammation occurs in subchondral bone seen in T2-weighted MRI as increase in signal density. Patients are treated initially by pain management. In patients who don't response to first line treatment invasive treatment like total knee replacement is done. The investigators designed this clinical study with the aim of evaluating therapeutic effects of intra-articular injection of bone marrow mesenchymal stem cells (BM-MSCs) in patients with severe knee osteoarthritis.

DETAILED DESCRIPTION:
This is single center, randomized, triple blind phase II clinical study. Patients will be divided into two groups of case and control. All subjects will undergo bone marrow aspiration. Mesenchymal stem cells will be isolated from bone marrow, cultured and transplanted back to the knee joint. Patients of case group will receive cell injection 1 and 4 months after bone marrow aspiration. Placebo will be administered in this group 6 months after the first injection. Patients of control group will receive placebo 1 and 4 months after bone marrow aspiration. They all receive cell injection 6 months after first placebo injection. Follow up visit will occur at 2 and 6 weeks, and 3 and 6 months after the first injection. Radiological exams will be performed before and 6 months after the first injection by MRI. Clinical quantitative assessment will measure joint function by the WOMAC index and pain by the visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis diagnosed by MRI

Exclusion Criteria:

* Pregnancy or lactating
* Positive tests for HIV, HCV, HBV
* Active neurologic disorder
* End organ damage
* Uncontrolled endocrine disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
physical function improvement | 2weeks
  Evaluation the physical function improvement Measured by WOMAC osteoarthritis index after cell injection.
change in pain density | 2 weeks
  Evaluation the changing of pain density measured by Visual Analogue Scale after cell injection.

SECONDARY OUTCOMES:
joint swelling | 3months
  Evaluation the joint swelling by physical examination after intra articular cell injection.
joint erythema | 3months
  Evaluation the joint erythem by physical examination after cell injection
deterioration of joint function | 3months
  Evaluation the deterioration of joint function by physical examination after intra articular cell injection.
Allergic reactions | 3months
  Evaluation the allergic reactions like skin rash,skin erythema,dyspenea by physical examination after cell injection

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Royan Cell therapy Center; Mohsen Emadeddin, MD, Principal Investigator — scientist
Locations (1):
- Royan Institute, Tehran, Iran